CLINICAL TRIAL: NCT06637540
Title: Clinical Validation of a Novel Ultrasound Probe (RescueDoppler) During Physiological Perturbations and Initiation Of- and Weaning from Cardiopulmonary Bypass in Adult, Cardiac Surgery Patients
Brief Title: Clinical Validation of a Novel Handsfree Doppler Ultrasound Device, RescueDoppler, in Adult Cardiac Surgery Patients
Acronym: RD_CPB
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: St. Olavs Hospital (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Other
Other Study IDs: 656036; CIV-NO-23-10-04 (Other: Norwegian Medical Products Agency)
Record Dates: First submitted 2024-10-03; First posted 2024-10-15 (Actual); Last update posted 2024-11-04 (Actual); Status verified 2024-09

CONDITIONS: Cardio-pulmonary Bypass; AORTIC VALVE DISEASES; Coronary Arterial Disease (CAD); Aortic Aneurysm of the Proximal Arch
Keywords: Handsfree Doppler Ultrasound; RescueDoppler; Pulsed wave Doppler Ultrasound; Cardiopulmonary bypass; Continous blood flow velocities in Cardiopulmonary bypass
MeSH Terms: conditions — Aortic Valve Disease

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (1):
- RescueDoppler patch with probe is attached to patients undergoing cardiac surgery. (Experimental): The RescueDoppler probe and patch are placed on the left side of the patient's neck in both preoperative and during surgery settings. The RescueDoppler system is connected to a screen with real-time bloodflow monitoring. The the blood flow curves are blinded for other health personell. After the cardiac surgery, the velocity curves are processed by the research team and synchronized with hemodynamic and respiratory data for analysis.
  Interventions: Device: RescueDoppler

INTERVENTIONS:
Device: RescueDoppler — Continous handsfree pulsed wave Doppler of the common carotid artery during cardiac surgery
  Other Names: RD; Carotid Pulsed waved Doppler; Carotid Doppler; Continous Carotid Doppler
Device: RescueDoppler — Continuous hands-free Doppler ultrasound of the common carotid artery during cardiac surgery
  Other Names: Rescue

SUMMARY:
The goal of this study is to evaluate a new device called RescueDoppler (RD), which measures continuous blood flow in the common carotid artery. The device is handsfree and operator- independent. The research will involve adult participants who are undergoing cardiac surgery at St. Olavs Hospital in Trondheim, Norway.

The aim of the first part of the study is to evaluate the RescueDoppler system in comparison to conventional Doppler ultrasound, which is commonly used to assess blood flow in carotid artery. The researchers will measure blood flow in the left common carotid artery in three different reversible situations:

* when the participant is resting,
* when there is increased blood flow (passive leg raise) and
* when there is decreased blood flow ( breathing against a resistance). We will initially conduct the investigation using the conventional Doppler. Subsequently, we will repeat the interventions with the RD patch positioned over the left common carotid artery.

The RD patch will stay positioned over the left carotid artery after the completion of the comparison phase. In the subsequent phase, the focus will shift to transitions between normal blood flow and low or absent blood flow and the RescueDopplers ability to detect. During cardiac surgery, participants will experience fluctuations in blood pressure, pulse, and circulation. By measuring blood flow with the RescueDoppler during these variations, researchers will evaluate the device´s capability to monitor different blood flow patterns.

Overall, the study aims to provide valuable insights into the effectiveness of the RescueDoppler in a clinical setting where changes in blood flow are expected.

DETAILED DESCRIPTION:
During high- risk surgery and critical illness, the main goal is to maintain an adequate cardiac output and oxygen delivery to vital organs. Accurate hemodynamic monitoring is essential in current critical care medicine and high-risk surgery. A systematic review and meta- analysis of non-invasive techniques compared to thermodilution as the reference standard, revealed only modest agreement and inadequate percentage error despite advances in medical technology over the last decades. This highlights the urgent need for reliable non-invasive method to monitor the perfusion of vulnerable organs during hemodynamically unstable situations.

During cardiac arrest (CA), the quality of cardiopulmonary resuscitation (CPR) relies on adequate chest-compressions and early shock when indicated. As such, the recommendations in international and European CPR guidelines consist of several methods to assess the quality of CPR. The pulse has been one of the most important diagnostic signs, first described in ancient medicine. Puls-check is still one of the recommended methods to guide CPR and evaluate possible return of spontaneous circulation (ROSC). However, the pulse-check is imprecise. In one study, 10% of healthcare workers detected pulse when the patient had cardiac arrest and only 45% were able to palpate pulse when the systolic blood pressure was higher than 80 mmHg. In addition, pulse check does not predict the magnitude of blood flow. In patients with out-of-hospital cardiac arrest (OHCA), a correlation has been shown between high end tidal carbondioxide (EtCO2) values during CPR and ROSC, as well as improved long-term survival. This method is recommended in international CPR guidelines as a decision-making tool to confirm the correct placement of the endotracheal tube in the trachea, serve as a quality indicator of CPR, and detect the return of a pulsatile heart rhythm. However, despite its utility, this method has known limitations in identifying ROSC and blood flow, and it has limited capacity to differentiate between various causes of cardiac arrest.

In cardiac surgery, particularly during cardiopulmonary bypass (CPB), patients experience various manipulations and circulatory changes that increase their vulnerability to complications in multiple organs. CPB is an extracorporeal technique that diverts the patient's blood away from the heart and lungs, rerouting it outside the body. This method replaces the normal physiological functions of the lungs and heart by managing oxygenation, ventilation, and maintaining adequate blood flow through several components of the CPB machine, including the pump, oxygenator (for gas exchange), tubing, and heat exchange units. The CPB pump functions like an artificial heart, generating continuous blood flow through a propeller mechanism. Blood is collected from the right heart or the vena cava (superior and/or inferior) and is then fully oxygenated before being returned via a cannula into the ascending aorta.

At St. Olavs Hospital, Trondheim University Hospital, the routine practice involves cross-clamping the ascending aorta and administering a cardioplegia solution-a cold fluid enriched with electrolytes and medication-to induce cardiac electromechanical silence during procedures. These physiological hemodynamic changes are of significant interest to the study group, as they involve transitions in blood flow from pulsatile (with a fully functioning heart) to non-pulsatile (due to cross-clamping and cardiac electromechanical silence) during the initiation of CPB, and back to pulsatile during weaning. While cerebral perfusion during CPB has been assessed in previous studies, to our knowledge, no prior research has specifically investigated cerebral blood flow during the initiation and weaning phases of CPB.

Protocols for hemodynamic management during CPB aim for a target flow of 2.2-2.8 liters/min/m², which approximates normal physiological values. It is recommended to monitor this flow based on oxygenation and metabolic parameters, including central venous oxygenation (SvO2), oxygen extraction (O2ER), Near-Infrared Spectroscopy (NIRS), venous carbon dioxide (VCO2), and lactate levels.

Critical illness and intensive care medicine involve a variety of medical conditions, making tailored monitoring challenging. Many available monitoring tools are invasive, require advanced equipment (such as PICCO and pulmonary artery catheters), or involve time-consuming interventions like passive leg raises, which may lead to the omission of hemodynamic guidance in busy clinical settings.

Ultrasound has emerged as a vital diagnostic and decision-making tool in critical care, particularly echocardiography, which can assess cardiac activity and function. However, it is user-dependent, requires specialized knowledge, and provides only a snapshot of the clinical situation.

The brain is particularly sensitive to hypoxia, and during cardiac arrest or surgery, hypoperfusion and vasoplegia can impair oxygen delivery, affecting treatment outcomes. Near-Infrared Spectroscopy (NIRS) is used to monitor oxygen delivery to the frontal brain during cardiac surgery, offering feedback to the treatment team on when to adjust hemodynamic support. Research indicates that a 20% decrease in regional hemoglobin oxygen saturation (rSO2) increases the risk of neurological complications.

Monitoring cerebral blood flow in the middle cerebral artery (MCA) with Transcranial Doppler (TCD) provides real-time data on blood flow during surgery. A significant reduction in MCA blood flow can signal complications, allowing for timely intervention to prevent brain ischemia. However, TCD requires ultrasound expertise and may present challenges in identifying the insonating window.

Carotid Doppler Ultrasound (CD) is an important method for monitoring blood flow and diagnosing carotid artery stenosis. Recently, it has been explored as a non-invasive hemodynamic monitoring tool. While some studies show promising results, the current literature presents mixed findings due to variations in patient populations and study designs. Like other ultrasound techniques, CD is user-dependent and offers only a snapshot of the situation.

In all the clinical situations mentioned, a precise, non-operator-dependent tool for continuous monitoring to guide and tailor treatment would be highly valuable. RescueDoppler is a novel Doppler ultrasound device designed to continuously measure blood flow in the common carotid artery. The concept originated from the need for improved methods to guide cardiopulmonary resuscitation (CPR) and monitor blood flow across various cardiac rhythms.

With the increasing body of research supporting carotid Doppler ultrasound as a non-invasive hemodynamic monitoring tool, the RescueDoppler technique becomes even more compelling. It is user-independent, featuring a self-adhesive patch that can be easily positioned using clear anatomical landmarks on the neck. While animal studies in cardiac arrest piglets show promising results, and unpublished data from a study of RD in in-hopsital and out-of-hospital cardiac arrest show that the RescuDoppler device is feasible. More human studies are still needed.

The overall aim of the study is to evaluate the RescueDoppler system's performance as a circulatory monitoring tool beyond feasability in patients going through different hemodynamic changes in a safe, clinical setting for better patient outcome. We will investigate subjects, aged 18-80, male and female, accepted for cardiac surgery either with coronary artery disease and/or valve or aortic disease at St. Olav´s Hospital, Trondheim, Norway. This is a single-center clinical study. We will include 42 patients. The enrollment periode will be Q1-Q4 2024. There will be no randomization or blinding in this study.

The two phases of the investigation will be conducted sequentially.

The primary investigation will compare and by that validate the RescueDoppler device against conventional Doppler ultrasound (CD). Blood flow velocities in the left common carotid artery will be measured first using CD, followed by the RD. The primary objective is to evaluate if the RescueDoppler device is noninferior to CD, by comparing the flow patterns and velocities recorded with the two methods. The primary endpoint is peak systolic velocity, secondary outcomes are diastolic velocity, time-averaged blood flow velocity (TAV) among others.

During cardiac surgery and CPB, the RescueDoppler patch will remain positioned over the left carotid artery. We will measure blood flow during key phases such as initiation of CPB, aortic cross-clamping, and weaning from CPB, and compare these measurements with hemodynamic and respiratory variables. The primary objective of this part is to evaluate the blood flow signals recorded continuously by the RescueDoppler device by assessing in subjects undergoing circulatory changes from pulsatile- to non-pulsatile blood flow when initiating- and back when weaning from CPB. The primary endpoint is time-averaged blood flow velocity (TAV).

Within the study, data about signal quality, fastening device functionality, data signal management and usefulness of blood flow information will be collected. Additionally, data will be collected to evaluate the initial clinical safety as per intended use.

ELIGIBILITY:
Inclusion Criteria:

1. Accepted for cardiac-, valve- and aortic surgery
2. Circulatory stable
3. Male and female
4. any BMI
5. Age 18-80

Exclusion Criteria:

1. Significant left carotid artery stenosis (> 50%)
2. Carotid stent or has had surgery to the left carotid artery
3. Emergency surgery
4. Hemodynamic unstable

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 42 (Actual)
Dates: Start 2024-01-28 (Actual); Primary Completion 2024-11-01 (Actual); Study Completion 2024-11-01 (Actual)

PRIMARY OUTCOMES:
Assessment of the velocity- time integral (the area under the blood flow curve in cm) at 25%, 50% and 75% decrease/increase in pulsatile blood flow. | From enrolment to the end after 11 months
  The primary objective is to assess the continuous blood flow signals in the left common carotid artery measured by the RescueDoppler device in a clinical setting in subjects undergoing planned circulatory changes from pulsatile- to non-pulsatile blood flow when initiating- and back when weaning from CPB. The primary endpoint as described in the Title.
Limits of agreement between peak systolic velocity (PSV in cm/sec) between conventional Doppler Ultrasound and RescueDoppler | From enrolment to the end after 11 months
  The objective is to evaluate if the RescueDoppler is noninferior to conventional Doppler ultrasound by comparing flow pattern and velocities by the two methods.

SECONDARY OUTCOMES:
Peak systolic velocity (PSV) in cm/s in correlation to a 25%,50%, 75% and 100% decrease/increase in pulsatile blood flow | From enrolment to the end after 11 months
The correlation between VTI and pulse pressure | From enrolment to the end after 11 months
  During CPB initiation and weaning
The correlation between PSV in cm/s and pulse pressure | From enrolment to the end after 11 months
The velocity time integral (VTI) | From enrolment to the end after 11 months
  The relationship between VTI in both CD and RD
Systolic and diastolic velocities in cm/s | From enrolment to the end after 11 months
  The realtionship between measurements in both CD and RD
Pulsatile index (PI) | From enrolment to the end after 11 months
  Compare the PI between conventional Doppler ultrasound and RescueDoppler Study the PI during initiation and weaning from CPB
Incidence of Treatment-Emergent Adverse Events | From enrolment to the end after 11 months
  Skin related adverse advents to RescueDoppler patch, -plaster,- hydrogel

CONTACTS AND LOCATIONS:
Locations (3):
- Norway (3):
  - St. Oalvs Hospital, Trondheim University Hospital, Trondheim
  - St.Olavs Hospital, Trondheim University Hospital, Trondheim
  - St. Olavs Hospital, Trondheim University Hospital, Trondheim

IPD SHARING:
Plan to Share IPD: Yes
ECG, invasive blood pressures, central venous pressure, blood flow velocities from both conventional ultrasound and the IMD.
Supporting Information: ICF, CSR
Time Frame: Starting 6 months after the publication of results and ending 2 years later
Access Criteria: A data sharing agreement must be signed and submitted to the steering committee, which includes the Principal Investigator (PI), Sponsor and Site Investigator (SI) from the hospital in the study.
URL: https://www.rescuedoppler.com

REFERENCES:
- [Background] Moritz S, Kasprzak P, Arlt M, Taeger K, Metz C. Accuracy of cerebral monitoring in detecting cerebral ischemia during carotid endarterectomy: a comparison of transcranial Doppler sonography, near-infrared spectroscopy, stump pressure, and somatosensory evoked potentials. Anesthesiology. 2007 Oct;107(4):563-9. doi: 10.1097/01.anes.0000281894.69422.ff. PMID 17893451
- [Background] Kamenskaya O, Klinkova A, Loginova I, Lomivorotov VV, Shmyrev V, Chernyavskiy A. Brain Oxygen Supply in Older Adults During Coronary Artery Bypass Grafting. J Cardiothorac Vasc Anesth. 2020 Dec;34(12):3275-3281. doi: 10.1053/j.jvca.2020.04.053. Epub 2020 May 14. PMID 32532692
- [Background] Adedipe AA, Fly DL, Schwitz SD, Jorgenson DB, Duric H, Sayre MR, Nichol G. Carotid Doppler blood flow measurement during cardiopulmonary resuscitation is feasible: A first in man study. Resuscitation. 2015 Nov;96:121-5. doi: 10.1016/j.resuscitation.2015.07.024. Epub 2015 Jul 30. PMID 26234896
- [Background] Gaspari R, Weekes A, Adhikari S, Noble V, Nomura JT, Theodoro D, Woo M, Atkinson P, Blehar D, Brown S, Caffery T, Douglass E, Fraser J, Haines C, Lam S, Lanspa M, Lewis M, Liebmann O, Limkakeng A, Lopez F, Platz E, Mendoza M, Minnigan H, Moore C, Novik J, Rang L, Scruggs W, Raio C. A retrospective study of pulseless electrical activity, bedside ultrasound identifies interventions during resuscitation associated with improved survival to hospital admission. A REASON Study. Resuscitation. 2017 Nov;120:103-107. doi: 10.1016/j.resuscitation.2017.09.008. Epub 2017 Sep 13. PMID 28916478
- [Background] Murkin JM, Adams SJ, Novick RJ, Quantz M, Bainbridge D, Iglesias I, Cleland A, Schaefer B, Irwin B, Fox S. Monitoring brain oxygen saturation during coronary bypass surgery: a randomized, prospective study. Anesth Analg. 2007 Jan;104(1):51-8. doi: 10.1213/01.ane.0000246814.29362.f4. PMID 17179242
- [Background] Rudolph JL, Sorond FA, Pochay VE, Haime M, Treanor P, Crittenden MD, Babikian VL. Cerebral hemodynamics during coronary artery bypass graft surgery: the effect of carotid stenosis. Ultrasound Med Biol. 2009 Aug;35(8):1235-41. doi: 10.1016/j.ultrasmedbio.2009.04.008. Epub 2009 Jun 21. PMID 19540657
- [Background] Lewis C, Parulkar SD, Bebawy J, Sherwani S, Hogue CW. Cerebral Neuromonitoring During Cardiac Surgery: A Critical Appraisal With an Emphasis on Near-Infrared Spectroscopy. J Cardiothorac Vasc Anesth. 2018 Oct;32(5):2313-2322. doi: 10.1053/j.jvca.2018.03.032. Epub 2018 Mar 20. PMID 30100271
- [Background] Baldi E, Caputo ML, Klersy C, Benvenuti C, Contri E, Palo A, Primi R, Cresta R, Compagnoni S, Cianella R, Burkart R, De Ferrari GM, Auricchio A, Savastano S. End-tidal carbon dioxide (ETCO2) at intubation and its increase after 10 minutes resuscitation predicts survival with good neurological outcome in out-of-hospital cardiac arrest patients. Resuscitation. 2022 Dec;181:197-207. doi: 10.1016/j.resuscitation.2022.09.015. Epub 2022 Sep 24. PMID 36162612
- [Background] Lomivorotov VV, Efremov SM, Kirov MY, Fominskiy EV, Karaskov AM. Low-Cardiac-Output Syndrome After Cardiac Surgery. J Cardiothorac Vasc Anesth. 2017 Feb;31(1):291-308. doi: 10.1053/j.jvca.2016.05.029. Epub 2016 Jul 29. No abstract available. PMID 27671216
- [Background] Polzl L, Thielmann M, Cymorek S, Nagele F, Hirsch J, Graber M, Sappler N, Eder J, Staggl S, Theurl F, Abfalterer H, Reinstadler SJ, Holfeld J, Griesmacher A, Ulmer H, Grimm M, Bauer A, Ruttmann-Ulmer E, Ruhparwar A, Bonaros N, Gollmann-Tepekoylu C. Impact of myocardial injury after coronary artery bypass grafting on long-term prognosis. Eur Heart J. 2022 Jul 1;43(25):2407-2417. doi: 10.1093/eurheartj/ehac054. PMID 35139192
- [Background] Anyanwu AC, Filsoufi F, Salzberg SP, Bronster DJ, Adams DH. Epidemiology of stroke after cardiac surgery in the current era. J Thorac Cardiovasc Surg. 2007 Nov;134(5):1121-7. doi: 10.1016/j.jtcvs.2007.06.031. PMID 17976438
- [Background] Eberle B, Dick WF, Schneider T, Wisser G, Doetsch S, Tzanova I. Checking the carotid pulse check: diagnostic accuracy of first responders in patients with and without a pulse. Resuscitation. 1996 Dec;33(2):107-16. doi: 10.1016/s0300-9572(96)01016-7. PMID 9025126
- [Background] Moule P. Checking the carotid pulse: diagnostic accuracy in students of the healthcare professions. Resuscitation. 2000 May;44(3):195-201. doi: 10.1016/s0300-9572(00)00139-8. PMID 10825620
- [Background] Soar J, Bottiger BW, Carli P, Couper K, Deakin CD, Djarv T, Lott C, Olasveengen T, Paal P, Pellis T, Perkins GD, Sandroni C, Nolan JP. European Resuscitation Council Guidelines 2021: Adult advanced life support. Resuscitation. 2021 Apr;161:115-151. doi: 10.1016/j.resuscitation.2021.02.010. Epub 2021 Mar 24. PMID 33773825
- [Background] Suriani I, van Houte J, de Boer EC, van Knippenberg L, Manzari S, Mischi M, Bouwman RA. Carotid Doppler ultrasound for non-invasive haemodynamic monitoring: a narrative review. Physiol Meas. 2023 Mar 1;43(10). doi: 10.1088/1361-6579/ac96cb. PMID 36179705
- [Background] van Houte J, Mooi FJ, Montenij LJ, Meijs LPB, Suriani I, Conjaerts BCM, Houterman S, Bouwman AR. Correlation of Carotid Doppler Blood Flow With Invasive Cardiac Output Measurements in Cardiac Surgery Patients. J Cardiothorac Vasc Anesth. 2022 Apr;36(4):1081-1091. doi: 10.1053/j.jvca.2021.09.043. Epub 2021 Oct 5. PMID 34756675
- [Background] Faldaas BO, Nielsen EW, Storm BS, Lappegard KT, Nilsen BA, Kiss G, Skogvoll E, Torp H, Ingul CB. Real-time feedback on chest compression efficacy by hands-free carotid Doppler in a porcine model. Resusc Plus. 2024 Feb 20;18:100583. doi: 10.1016/j.resplu.2024.100583. eCollection 2024 Jun. PMID 38404755
- [Background] Faldaas BO, Nielsen EW, Storm BS, Lappegard KT, How OJ, Nilsen BA, Kiss G, Skogvoll E, Torp H, Ingul C. Hands-free continuous carotid Doppler ultrasound for detection of the pulse during cardiac arrest in a porcine model. Resusc Plus. 2023 Jun 20;15:100412. doi: 10.1016/j.resplu.2023.100412. eCollection 2023 Sep. PMID 37448689
- See also: Related Info — http://rescuedoppler.com